CLINICAL TRIAL: NCT04608526
Title: Evaluation of the Relationship Between Tooth Decay and Trabecular Bone Structure in Pediatric Patients by Fractal Analysis Method: A Retrospective Study
Brief Title: Relationship Between Tooth Decay and Trabecular Bone
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Sema Aydınoglu, assistant professor, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 2020/127
Record Dates: First submitted 2020-10-20; First posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Dental Caries in Children; Pediatric Patients; Radiology
Keywords: Disturbances in dental development; fractal analysis; pediatric patients; radiology

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Patients without deep dentin caries / apical rarefying osteitis
  Interventions: Diagnostic Test: Fractal analysis
- Group 2: Patients with deep dentin caries / apical rarefying osteitis on the right or left sides
  Interventions: Diagnostic Test: Fractal analysis
- Group 3: Patients with deep dentin caries / apical rarefying osteitis on either the right and left side
  Interventions: Diagnostic Test: Fractal analysis

INTERVENTIONS:
Diagnostic Test: Fractal analysis — Fractal dimension (FD) analysis, which can be measured in panoramic radiographs, is a technique that can be used to measure mandibular trabecular architecture and to determine early periodontal changes in alveolar bone. Fractal analysis method, which has become more and more popular in recent years; has features such as being easily accessible, not being affected by variables such as projection geometry and radiological density and providing objective data about trabecular structures. It can be measured in the patients' existing panoramic images and does not require extra imaging and material.

SUMMARY:
Chewing, a movement that matures with experiences, has effects on the growth and development of the stomatognathic system. Tooth decay, which is known to have effects on chewing, can affect the jaw bone due to its indirect effect on the mechanical forces transmitted to the jaw bone. This study was aimed to evaluate the relationship between dental caries and jaw bone trabeculation during the growth and development processes in children by fractal dimension analysis method. 40 patients with deep-dentin caries / apical rarefying osteitis on the right or left side, 40 patients with deep-dentin caries / apical rarefying osteitis on either the right and left sides and 40 patients without deep-dentin caries / apical rarefying osteitis between 8-13 ages were randomly selected. Digital panoramic images of the selected patients were analyzed with fractal dimension analysis.

ELIGIBILITY:
Inclusion Criteria:

* Panoramic radiographs of systemically healthy 8-13 years-old patients,
* Who applied to the Clinic between January 2018 and April 2020 were retrospectively scanned.
* Patients with 1st molars whose root development was completed and the 2nd molars not erupted yet were included.

Exclusion Criteria:

* Patients with temporomandibular joint disorders, any systemic disease, exposed to trauma in the area to be measured, received orthodontic treatment for the last 2 years or had an ongoing orthodontic treatment, unilateral / bilateral cross-bite and had parafunctional habits in their anamnesis were excluded.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: * systemically healthy,
  * 8-13 years-old,
  * applied to the Clinic between January 2018 and April 2020 patients
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-10-19 (Actual)

PRIMARY OUTCOMES:
The effects of dental caries on the jawbone in children aged between 8-13 years | for two months from the beginning of the study
  Digital panoramic radiographs of the patients included in the study were recorded in high resolution TIF (tagged image file) format to ensure standardization of the images and adjusted to 2836 x 1500 pixels. ImageJ version 1.53a, and bundled with 64-bit Java for Windows (National Institutes of Health, Bethesda) were used for fractal analysis of the images.
  Fractal analysis on digital panoramic radiographs transferred to ImageJ (National Institutes of Health, Bethesda) program, 3 ROI (region of interest) areas of 15x15 pixels were determined for each patient with condyle, antegonial notch in the right and left hemimandible and in the center of the ramus.The number of frames containing the trabecular structure and the total number of frames were calculated for different dimensions. The values were transferred to the logarithmic scale and the slope of the curve fitting the points on the graph gave the result of the fractal measurement.

CONTACTS AND LOCATIONS:
Overall Officials: SEMA AYDINOĞLU, Study Director — Recep Tayyip Erdogan University Training and Research Hospital
Locations (1):
- Sema Aydinoğlu, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No